CLINICAL TRIAL: NCT05104359
Title: Should COVID-19 Quantitative Antibody Titers be Implemented to Guide COVID-19 Booster Vaccinations Regardless of HIV Status, Immunosuppression, or Age?
Brief Title: COVID-19 Quantitative Antibody Titers & Booster Vaccinations
Status: Completed | Type: Observational
Sponsor: Epividian (Industry)
Collaborators: AIDS Healthcare Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: COL2021-001
Record Dates: First submitted 2021-11-01; First posted 2021-11-03 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; COVID-19 Vaccines; Immunogenicity, Vaccine
Keywords: COVID-19; Observational; Vaccination; Antibody; Booster
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational — HIV-positive versus HIV-negative patients, individuals with at least 2 measurements of antibody levels, and boosted individuals are the subgroups of interest.

SUMMARY:
This is an observational study aiming at describing COVID-19 vaccination outcomes among HIV-positive and HIV-negative individuals, using electronic health records to observe their usual clinical care. This study will describe levels of COVID-19 vaccine response (i.e., Ig spike antibody measurements). Rates of antibody level decay after vaccination will be assessed. The efficacy of using antibody levels to help guide the timing of booster doses among HIV-negative and HIV-positive patients will be evaluated.

DETAILED DESCRIPTION:
The aim of this study is to assess levels of COVID-19 vaccine response through measuring surrogate Ig spike antibody measurements, to determine the rates of antibody level decay after vaccination, and to measure the efficacy of utilizing these antibody measurements to help guide the timing of booster doses among HIV-negative and HIV-positive patients.

The study population will include adults who were fully vaccinated against SARS-CoV-2 virus (i.e., two doses of Pfizer or Moderna vaccines or one dose of the J&J vaccine), and have received a Roche SARS-CoV-2 Semi-Quant Spike Ig Ab test at least 3 weeks after full vaccination as part of their usual clinical care at AHF Midtown Manhattan Healthcare Center.

Incidence rates of COVID vaccine response levels (i.e., adequate, low, non-response) will be estimated using univariate Poisson regression, overall and by vaccine type. Among individuals with at least two antibody measurements, rates of antibody levels decay will be estimated using univariate linear regression, overall and stratified by HIV status, vaccine type and baseline CD4 cell count. In the sub-population of individuals who received a COVID vaccine booster, vaccination and antibody response will be characterized at least 3 weeks after the booster is received. Univariate linear regression will be used to estimate rates of antibody levels decay, among individuals with at least two antibody measurements, including one after the booster dose. Rates of response decay will be produced overall, and stratified by HIV status, booster type and baseline CD4 cell count.

ELIGIBILITY:
Inclusion Criteria:

* Cared for at AHF Midtown Manhattan Healthcare Center and followed in the OPERA observational database
* Active in care in the last 24 months
* Fully vaccinated against SARS-CoV-2 virus, implemented as 21 days after the second Pfizer or Moderna injections, 21 days after the one J&J injection
* Received a Roche SARS-CoV-2 Semi-Quant Spike Ig AB test after full vaccination as usual clinical care

Exclusion Criteria:

* Unvaccinated or partially vaccinated against SARS-CoV-2 virus
* Never tested with a SARS-CoV-2 Semi-Quant Total AB test after full vaccination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals presenting for care at AHF Midtown Manhattan Healthcare Center who received COVID-19 vaccination and antibody testing; followed through their electronic health records in the OPERA Observational Database.
Sampling Method: Non-Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Vaccine Response | >21 days
  Levels of Roche SARS-CoV-2 Semi-Quant Spike Ig antibody

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Hsu, MD, Principal Investigator — AHF Midtown Manhattan
Locations (1):
- AHD Manhattan Midtown HCC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT05104359/Prot_SAP_000.pdf